CLINICAL TRIAL: NCT05831683
Title: Standard Operating Procedure As a Valuable Tool to Increase Adherence to Lung Protective Ventilation Among Anesthesiologists.
Status: Completed | Type: Observational
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Michal Kalina, Principal investigator, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Other Study IDs: SOP LPV study
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Adherence, Treatment
Keywords: Lung Protective Ventilation; Ventilation; Standard Operating Procedure; Adherence; Mechanical Ventilation
MeSH Terms: conditions — Treatment Adherence and Compliance; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A - Current state: In this group, ventilator parameters will be recorded before the SOP introduction. We will analyze PEEP, Pplat, driving pressure, VT/IBW, and the number and phase of recruitment maneuvers during general anesthesia.
- Group B - After SOP introduction: In this group, ventilator parameters will be collected after the SOP introduction. We will analyze PEEP, Pplat, driving pressure, VT/IBW, and the number and phase of recruitment maneuvers during general anesthesia.
  Interventions: Other: Introduction of Standard Operating Procedure regarding lung protective ventilation during general anaesthesia.

INTERVENTIONS:
Other: Introduction of Standard Operating Procedure regarding lung protective ventilation during general anaesthesia. — The Standard Operating Procedure document will be introduced. The SOP document will cover the theoretical background, definition, and recommendations/criteria of LPV. The SOP document will reflect the most recent LPV guidelines.
  Groups: Group B - After SOP introduction

SUMMARY:
Lung Protective Ventilation (LPV) is considered the gold standard of care nowadays. Even though, all over the world reported adherence to this concept, among anesthesiologists, is only 15%. The investigators hypothesized that the introduction of the Standard Operating Procedure (SOP) document will increase adherence to LPV among anesthesiologists. In this study, the investigators will record ventilating parameters during general anesthesia using Care Station Insights software. Then, the investigators will evaluate the recorded parameters and match them with LPV criteria. The adherence level to every parameter separately will be counted in percentage.

DETAILED DESCRIPTION:
In this study, the investigators will start by stating the current adherence level to the LPV concept during general anesthesia among anesthesiologists. Adherence will be calculated as percentage of cases that will met the criteria. The evaluation will be based on saved data in Care Station Insights software from General Electric. This software is running on anesthesia machines GE Aysis CS2.

The investigators will record and evaluate:

* Positive End Expiratory Pressure (PEEP) [cmH2O]
* Plateau Pressure (Pplat) [cmH2O]
* driving pressure [cmH2O]
* Tidal Volume/Ideal Body Weight (VT/IBW)
* number of recruitment maneuvers during a case
* phase of a case when recruitment maneuver is done (induction/maintenance/emergence)

Each parameter will be evaluated separately. The adherence level for each parameter will be interpreted as a percentage of cases that meet the LPV criteria in terms of the given parameter. The investigators will evaluate the 100 most recent cases, before the SOP introduction, to state the current adherence level.

After stating the current adherence level to the LPV during general anesthesia, the investigators will introduce the Standard Operating Procedure document (SOP). SOP introduction will be supplemented with an educational program regarding LPV.

The SOP will include:

* the definition of LPV
* the theoretical background of LPV
* LPV strategy recommendations/criteria

The educational program:

* set of 11 half-hour-long sessions with LPV experts
* induction recommendations
* preoxygenation recommendations
* PEEP intraoperative recommendations
* LPV strategy during general anaesthesia and perioperative complications
* LPV in specific situations
* laparoscopy
* robotics surgery
* pronation
* recruitment maneuvers during general anaesthesia
* extubation recommendations
* neuromuscular blockade and monitoring recommendations
* Adequacy of Anaesthesia (AoA) strategy

Then, the investigators will begin with recording the second set of ventilatory parameters. The investigators will collect the very same parameters to state the current adherence level to LPV during general anesthesia as in the first data set. Ventilatory parameters will be collected the same way as for the first data set, with the use of Care Station Insights software. Anesthesiologists giving the anesthesia care will not know neither the goal of the study nor which parameters are recorded.

After finishing collecting the second data set, based on sample size calculation, the investigators will evaluate these. The evaluation process will be identical to the evaluation process of stating the current adherence level. The investigators will evaluate each parameter separately. Adherence for each parameter will be interpreted as a percentage of cases that meet the LPV criteria in terms of the given parameter.

At the finish, the investigators will compare adherence levels before and after the SOP introduction.

ELIGIBILITY:
Inclusion Criteria:

* A general anaesthesia case with the airway secured with the endotracheal tube

Exclusion Criteria:

* General anaesthesia without time cycled ventilator regime
* General anaesthesia without airway secured with an endotracheal tube
* General anaesthesia in which the care is given by a member of the study team of this study
* General anaesthesia in which one lung ventilation is used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventilatory parameters will be recorded during a case of general anesthesia with the use of an endotracheal tube and a time-cycled ventilatory regime. The recording will be from adult-only operating theatres.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
SOP increase adherence level to lung protective ventilation strategy | From initiation of mechanical ventilation till extubation, assessed up to 8 hours.
  The primary objective of the study is to demonstrate that the introduction of the SOP document regarding LPV during general anesthesia will increase adherence (number of cases that meet the SOP criteria) to the LPV concept during general anesthesia among anesthesiologists. We will collect ventilatory parameters during general anesthesia. These parameters will be then evaluated against LPV recommendations. The level of adherence will be counted as a percentage of cases that meets the LPV criteria. For each parameter, we will count the level of adherence separately.

SECONDARY OUTCOMES:
SOP increase the total number of recruitment maneuvers during a case | From initiation of mechanical ventilation till extubation, assessed up to 8 hours.
  The secondary aim of this study is to demonstrate that the introduction of the SOP document regarding LPV during general anesthesia will increase the total number of recruitment maneuvers. With the use of Care Station Insights software, we will record how many recruitment maneuvers are done during general anesthesia. We will compare the total number in the first data set (before the SOP introduction) and in the second data set (after the SOP introduction).
SOP increase the total number of recruitment maneuvers within the first ten minutes in a case. | From initiation of mechanical ventilation till extubation, assessed up to 8 hours.
  The secondary aim of this study is to demonstrate that the introduction of the SOP document regarding LPV during general anesthesia will increase the total number of recruitment maneuvers that are performed within the first ten minutes after securing the airway. We will count the number of recruitment maneuvers done within the first ten minutes and we will compare the count in the first data set (before the SOP introduction) and in the second data set (after the SOP introduction).
SOP increase the number of cases with PEEP greater than six cmH2O | From initiation of mechanical ventilation till extubation, assessed up to 8 hours.
  The secondary aim of this study is to demonstrate that the introduction of the SOP document regarding LPV during general anesthesia will result in a statistically significant increase in cases with a PEEP value greater than eight cmH2O. We will record the PEEP during a case. For evaluation, we will use the average value of PEEP during the case. We will compare the average PEEP in the first data set (before the SOP introduction) and in the second data set (after the SOP introduction).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kalina, MUDr., Principal Investigator — Krajská Zdravotní a.s. Klinika anesteziologie, perioperační a intenzivní medicíny MNUL a FZS UJEP
Locations (1):
- Masarykova Nemocnice v Ústí nad Labem, Krajská Zdravotní a.s., Ústí nad Labem, Ústí Nad Labem Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michal K, Jan B, Josef S, Patricia V, Adela B, Roman S, Vladimir C. The mandatory educational module increases the effect of implementing the standard operating procedure and adherence to the lung-protective ventilation concept during anaesthesia. BMC Med Educ. 2025 Oct 2;25(1):1333. doi: 10.1186/s12909-025-07923-z. PMID 41039371